CLINICAL TRIAL: NCT04232982
Title: The Role of Transscleral Cyclophotocoagulation in Patients Undergoing a Boston Keratoprosthesis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Fonds de recherche en ophtalmologie de l'Université de Montréal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CE19.253
Record Dates: First submitted 2020-01-13; First posted 2020-01-18 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Glaucoma; Eye Diseases; Cornea Disease
Keywords: Boston keratoprosthesis; Transscleral cyclophotocoagulation; Micropulse transscleral cyclophotocoagulation; G-Probe Transscleral cyclophotocoagulation
MeSH Terms: conditions — Glaucoma; Eye Diseases; Corneal Diseases

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, single blinded study with two interventional arms and one historical cohort as controls.
Who Masked: Participant
Masking Description: Patients will not be aware of which type of cyclophotocoagulation treatment they will be allocated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MicroPulse Treatment (Experimental): Prophylactic transscleral cyclophotocoagulation treatment, delivered by micropulse waves will be given 4-8 weeks before the Boston keratoprosthesis surgery.
  Interventions: Procedure: Transscleral cyclphophotocoagulation using the Micropulse system ( IRIDEX IQ810 Laser systems, Mountain View, CA).
- G-Probe Treatment (Experimental): Prophylactic transscleral cyclophotocoagulation treatment, delivered with a diode laser using the G-Probe device, will be given 4-8 weeks before the Boston keratoprosthesis surgery.
  Interventions: Procedure: G-Probe transscleral cyclphophotocoagulation (Iris Medical Instruments, Montain View, CA)
- Historical Cohort (No Intervention): An historical cohort composed of patients who received a Boston keratoprosthesis between january 2017 and january 2019 will be included. Only patients who did not receive any glaucoma treatment 3 months before their surgery will be included. A total of 10 patients will be selected with the goal of matching the preoperative characteristics of the interventional patients.
  This group will serve as the control group in our study. Retrospective chart review will be performed for this branch.

INTERVENTIONS:
Procedure: Transscleral cyclphophotocoagulation using the Micropulse system ( IRIDEX IQ810 Laser systems, Mountain View, CA). — Treatment will be applied over the limbal area to treat the ciliary body. The treatment will be delivered with an energy of 2000mW, a cycle of 31,33% and an on/off time of 0,5ms and 1,1ms. It will be delivered around a 360° surface with avoidance of the 3 and 9 o'clock areas. The treatment will be delivered during 80 secondes in each hemisphere and will be repeated twice, for a total of 320 secondes.
  Other Names: MP-TSCPC
  Arms: MicroPulse Treatment
Procedure: G-Probe transscleral cyclphophotocoagulation (Iris Medical Instruments, Montain View, CA) — Treatment will be applied over the limbal area to treat the ciliary body. Sixteen (16) shots in total, which is four (4) shorts per quadrants, will be transmitted with a power from 1750 to 2000mV (titrating according to an audible "pop") for a length of 2,0 secondes per shots. Treatment will be delivered around a 360° surface and avoiding the 3 and 9 o'clock areas.
  Arms: G-Probe Treatment

SUMMARY:
The Boston keratoprosthesis (KPro) is a special plastic device that is used to replace a sick cornea (transparent part of the eye, in front of the iris) in order to restore vision in patients who have failed traditional corneal transplants or have a very poor prognosis of success.

Glaucoma is a chronic disease which causes optic nerve damage secondary to high pressure inside the eye and could lead to vision loss in the long term. Glaucoma is highly prevalent in patients who require a KPro and even more after their procedure.

In order to decrease the intra-ocular pressure, surgeons can use multiple eyedrops. Unfortunately, following the KPro surgery, eyedrops lose their efficiency because they are less absorbed by the eye.

The transscleral cyclophotocoagulation (TS-CPC) is a laser treatment used in advanced refractory glaucoma. This laser helps decrease the intra-ocular pressure and have a better control of the disease. There are different methods of laser transmission, including the continuous transmission (G-Probe) and the micro-pulsation method (Micopulse). Given the high prevalence of glaucoma in patients receiving a KPro, the investigators are studying the effect of giving the TS-CPC treatment prophylactically to patients before their Boston keratoprosthesis.

Our hypothesis is that prophylactic TS-CPC will decrease glaucoma progression as well as the risks of developing glaucoma following the Boston keratoprosthesis .

METHOD The investigators aim to recruit twenty (20) patients who are scheduled to receive Boston KPro. Participants will be randomized into two groups: 1) Groupe 1 will receive a prophylactic treatment of transscleral cyclophotocoagulation a G-Probe. 2) Groupe 2 will receive a prophylactic treatment of transscleral cyclophotocoagulation with a micropulse transmission (MicroPulse). The patients will receive their laser treatment by a glaucoma specialist 4 to 8 weeks before their KPro surgery. One week following their laser treatment, the participants will be examined by their glaucoma specialist.

Following their KPro surgery, patients will have a follow-up at day-1, weeks 1 and 2, months 1 and 3, then every 4 to 6 months for 5 years. Additional non-invasive glaucoma tests will be performed twice during the first 3 months following the surgery and will be repeated every 4-6 months. Visual acuity results, the visual field tests and rates of post-operative complications will be compared between the different groups.

DETAILED DESCRIPTION:
RATIONAL OF THE STUDY

The Boston keratoprosthesis (KPro) type is an artificial cornea used to restore vision in patients who have failed traditional corneal transplants or have a poor prognosis of success. A number of innovations have improved the postoperative prognosis since its first creation. However, glaucoma is still one of the leading causes of significant vision loss following the surgery, despite the clarity of the anterior segment.

The prevalence of glaucoma in KPro candidates is highly elevated (36-76%). Indeed, pathologies requiring a Boston keratoprosthesis and history of previous ocular surgeries are themselves risk factors for glaucoma. Furthermore, the corneal opacity and irregularities lead to poor visualization of the optic nerve and incorrect intra-ocular pressure (IOP) measurements. Thus, the prevalence of glaucoma preoperatively is most likely underestimated.

Following the KPro, the increase of IOP or the new diagnosis of glaucoma is estimated between 8 and 35% per year. Additionally, the IOP cannot be determined by the traditional tonometry and is estimated by digital palpation. This leads to treatment follow-up being difficult and limited. For those reasons, it is suggested by experts to insert a glaucoma drainage device during the Boston keratoprosthesis surgery for all patients.

In perspective, the transscleral cyclophotocoagulation (TS-CPC) is one of the cyclodestructive procedures used for severe glaucoma. It leads to destruction of the ciliary body epithelium and reduction of aqueous humour production which can reduce the IOP.

Different transmission techniques are available and include the Micropulse diode laser (MP-TSCPC, IRIDEX IQ810 Laser systems, Mountain View, CA) and the semiconductor system with the G-Probe (IRIS Oculight SLx, IRIS Medical Inc., Mountain View, CA). These two systems differ by their transmission method, which is via pulsation waves (Micropulse) or continuous transmission (G-Probe).

In the literature, there are limited studies who have examined the role and the impact in the long term of the transscleral cyclophotocoagulation in patients receiving a Boston keratoprosthesis.

HYPOTHESIS Our hypothesis is that prophylactic transscleral cyclophotocoagulation will decrease glaucoma progression as well as the risks of developing glaucoma following the Boston keratoprothesis.

OBJECTIFS Our primary objective in this study is to examine if the use of prophylactic transscleral cyclophotocoagulation treatment with the G-Probe or the Micropulse (MP-TSCPC) methods prophylactically has a positive impact in the diagnosis of the progression of glaucoma in patients receiving a keratoprosthesis, without additional glaucoma surgery.

For more information on our primary and secondary criteria, please see in the below sections.

METHODS

Study design: This is a prospective, randomized, single blinded trial of patients receiving a KPro at the CHUM, with a historical cohort as a control group.

Recruitment: Patients will be recruited by their cornea surgeons, risks and benefits of the studies will be explained. An informed consent form will be obtained.

Prospective Branch of the Study

The study will include twenty (20) patients in the prospective branch of this study in the spam of two (2) years. Patients will receive a cyclophotocoagulation treatment 4-6 weeks before their Boston Keratoprosthesis surgery. Patients will be randomly assigned to either one of the TS-CPC treatment (Micro-Pulse or G-Probe).

Following the KPro surgery, if any additional glaucoma surgery is necessary (including the insertion of a glaucoma drainage device), these treatment options will be offered to the participants, as per standard of care.

For more information regarding the intervention's arms, see the section below.

Control group- cohort study

A control group composed of a historical cohort of ten (10) patients who did not receive any glaucoma surgery or TS-CPC 3 months before their Boston keratoprosthesis will be included in the historical cohort.

Indeed, when reviewing the literature, given the high prevalence of glaucoma in this population and the current recommendation of inserting a glaucoma drainage device (GDD) in patients receiving a KPro, it would be ethically non-acceptable to have a prospective group without any prophylactic treatment. Moreover, given the fact that we are going to compare between the different groups the need of additional glaucoma surgery, we cannot include a control group in which patients will receive a tube before or during their KPro surgery.

Follow-up

Patients will be followed by a glaucoma specialist 1 week following the TS-CPC treatment, as per standard of care.

After the Boston KPro, postoperative follow-up will be organized as per standard of care and will be similar across the three groups. Patients will be seen at postoperative day-1, weeks 1 and 2, months 1 and 3, then every 4 to 6 months for 5 years. During those visits, visual acuity as well as IOP and a complete slit-lamp exam will be performed. Furthermore, an optic nerve optical coherence tomography (OCT) will be performed and two visual fields test (SITA-Fast and Goldman) will be performed during the first and third month post-KPro. These particular tests will be repeated every 4-6 months, for a period of 5 years.

STATISTICAL ANALYSIS

Sample size

The investigators used the G-Power software to determine our sample size. Given that our primary endpoint is a continuous variable, the investigators used a student t-test with a power of 90%, an alpha of 0,05 and an effect size of 2,6. For the effect size, it was determined based of a difference clinically significant of 20% with the progression of the cup-to-disc ratio in KPro patients. Of note, this study only included the average and not the standard of deviation. The investigators assumed that the standard of deviation increases proportionally to the mean.

Statistical analysis Binary variable will be compared across the three groups using a chi square test. For continuous variable, such as the cup-to-disc ratio progression and the thinning of the Retinal Nerve Fiber Layer (RNFL), an ANOVA test will be performed. A test using an alpha parameter of 0,05 will be judged as clinically significant.

The visual acuity will be expressed in LogMar and its evolution will be compared across the three groups. The investigators will compare the rate of no light perception (NLP) between the three groups. Given that a previous study showed a 16% rate of NLP after 5 years. The investigators will consider a difference of 5% as clinically significant.

A Kaplan-Meir survival curve will be performed for: (1) the loss of light perception and (2) the need of a second intervention for glaucoma control. A Log-rank test will be performed to determine if those variables are statistically different across the groups.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients
* Able to give an informed consent
* Capable of being followed during the study
* Candidate for the Boston keratoprosthesis type I

Exclusion Criteria:

* Patients younger than 18 years old or older than 80 years old
* Unable to give an informed consent
* Participating to another interventional glaucoma study
* Patients who received a glaucoma surgery or procedure (glaucoma drainage device or TS-CPC treatment) 3 months before their initial visit.
* Unable to wear a therapeutic contact lens secondary to eyelid malformation
* Severe Ocular surface Disease with keratinization
* Intra-ocular tumor
* Terminal Glaucoma
* Phthisis bulbi
* Ocular albinism

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-01-30 (Actual); Primary Completion 2034-12-01 (Estimated); Study Completion 2036-12-01 (Estimated)

PRIMARY OUTCOMES:
Cup-to-disc ratio | 5 years
  Rate of progression of the optic nerve cup-to-disc ratio

SECONDARY OUTCOMES:
No light perception | 5 years
  Rate of patients with no light perception
Need of additional glaucoma intervention | 5 years
  Number of patients requiring any additional glaucoma surgery or procedure ( glaucoma drainage device, transscleral cyclophotocoagulation treatment etc.)
Goldman visual field loss of 30% or more. | 5 years
  Number of patients who lose more than 30% or more of their Goldman visual field during their follow-up. The first first two visual fields will be used at baseline as a baseline reference for comparaison.
Retinal Nerve Fiber Layer thinning | 5 years
  Percentage of patients with Retinal Nerve Fiber Layer thinning on Optical Coherence Tomography.

OTHER OUTCOMES:
Complications related to transscleral cyclophotocoagulation treatment | 5 years
  Rate of known complications of transscleral cyclophotocoagulation treatment (hypotony, phthisis bulbi)
Complications related to the Boston keratoprosthesis | 5 years
  Rate of known complications of the Boston keratoprosthesis (corneal melt, retroprosthetic membrane, retinal or choroid detachment)

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Claude Robert, MD, MSc, Principal Investigator — Ophthalmology Department, Centre Hospitalier de l'Université de Montreal
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Robert MC, Pomerleau V, Harissi-Dagher M. Complications associated with Boston keratoprosthesis type 1 and glaucoma drainage devices. Br J Ophthalmol. 2013 May;97(5):573-7. doi: 10.1136/bjophthalmol-2012-302770. Epub 2013 Feb 23. PMID 23435225
- [Background] Vajaranant TS, Liu J, Wilensky J, Cortina MS, Aref AA. Innovative approaches to glaucoma management of Boston keratoprosthesis type 1. Curr Ophthalmol Rep. 2016 Sep;4(3):147-153. doi: 10.1007/s40135-016-0102-3. Epub 2016 Jul 26. PMID 28529825
- [Background] Jabbour S, Harissi-Dagher M, Agoumi Y, Singh H, Robert MC. Cyclophotocoagulation in the Control of Glaucoma in Patients With the Boston Keratoprosthesis Type 1. Cornea. 2020 Feb;39(2):181-185. doi: 10.1097/ICO.0000000000002064. PMID 31335536
- [Background] Rivier D, Paula JS, Kim E, Dohlman CH, Grosskreutz CL. Glaucoma and keratoprosthesis surgery: role of adjunctive cyclophotocoagulation. J Glaucoma. 2009 Apr-May;18(4):321-4. doi: 10.1097/IJG.0b013e3181815485. PMID 19365199
- [Background] Patel S, Takusagawa H, Shen L, Dohlman C, Grosskreutz C. Long-term complications associated with glaucoma drainage devices and Boston keratoprosthesis. Am J Ophthalmol. 2012 Jul;154(1):207-8; author reply 208-9. doi: 10.1016/j.ajo.2012.02.033. No abstract available. PMID 22709836
- [Background] Crnej A, Paschalis EI, Salvador-Culla B, Tauber A, Drnovsek-Olup B, Shen LQ, Dohlman CH. Glaucoma progression and role of glaucoma surgery in patients with Boston keratoprosthesis. Cornea. 2014 Apr;33(4):349-54. doi: 10.1097/ICO.0000000000000067. PMID 24531120